CLINICAL TRIAL: NCT00774293
Title: Preliminary Study of a Homoeopathic Association in Patients Undergoing Aortic Valve Surgery.
Brief Title: Homoeopathic Association in Aortic Valve Surgery
Acronym: OMEO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BOIRON (Industry)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Philipe Belon, Boiron
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Boiron 041052
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Aortic Valve Replacement
Keywords: Homoeopathic treatment,; heart surgery,; randomized clinical trial
MeSH Terms: interventions — Arnicae flos extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Arnica 5CH and Bryonia 9CH (homeopathic drugs)
  Interventions: Drug: Arnica and Bryonia
- 2 (Placebo Comparator): placebo Arnica 5CH and Bryonia 9CH
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — 5 placebo granules for Arnica 5 CH and 5 placebo granules for Bryonia 5 CH
  Arms: 2
Drug: Arnica and Bryonia — Arnica 5CH granules, 5 per day plus Bryonia 5CH Granules, 5 per day for 5 days
  Arms: 1

SUMMARY:
Randomized, parallel group, placebo controlled study to assess the effect of an homoeopathic association of Arnica 5 CH et Bryonia 9 CH during aortic valve surgery with extra corporeal circulation, to alleviate inflammation, haemorrhage, myocardial ischemia and pain. This is a pilot study; a confirmative study will be set up if this study is positive.

The study treatment will start the day before surgery, and will comprise 5 granules of each homoeopathic medication, Arnica 5 CH and Bryonia 9 CH, or their matching placebo TID during 5 days, in addition to all routine treatments.) Two groups of 45 patients will be included. Patients have to be over 18 years, to undergo aortic valve surgery only, have no known allergy to one of the study drugs, sign a consent form, and must not have received anti inflammatory drug in the 3 days before surgery. The primary criteria include the amount of drained liquid from the chest, and the CRP evolution from baseline to the 7th postoperative day. Secondary criteria address inflammation, haemorrhage, ischaemia, and pain. A follow-up phone call is given to the patients 30 days after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, undergoing aortic valve surgery with extra corporeal circulation

Exclusion Criteria:

* acute infectious or inflammatory concomitant disease, known allergy to one of the investigational products, Patients who did not sign the study consent form, patients having received during the 3 days before surgery any corticoids or non steroid anti-inflammatory drug, patient undergoing a surgery other than surgery of the aortic valve in the same intervention, patient undergoing an iterative cardiac surgery, patients under 18 years, patient over 18 years under the protection of the law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-09; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Amount of drained liquid from the mediastinum or the pleura | At drain removal
plasma C reactive protein (CRP) at anaesthesia induction, plasma C reactive protein (CRP) | Day 2 and Day 7

SECONDARY OUTCOMES:
Evolution of body temperature from before surgery to day 2 after surgery. | Day 2
Time from the end of extra corporeal circulation to closure of the thorax, | Closure of thorax
Amount of transfusions of erythrocytes, platelets, plasma. | Day 7
Visual analogical scale (VAS) for pain every 6 hours during stay in PACU, and every day afterwards to day 7, | To day 7
Amount of analgesic drugs, paracetamol and morphine. | Day 7
EKG before surgery, 24 and 48 hours after surgery. | 48 hours
Plasma troponin I at induction of anaesthesia, 6, 24 and 48 hours after surgery. | 48 hours
Quality of cicatrisation of sternotomy immediately after surgery, at day 2 and 7 after surgery, on a 4 point scale. | Day 7
Clinical events: death, new surgery for haemostasis or infection within 2 weeks of surgery, and any event occurring within 30 days after surgery. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Lehot, MD, Principal Investigator — Hospices Civils de Lyon, Lyon, France
Locations (1):
- Anaesthesy service, Louis Pradel Hospital, Lyon, France